CLINICAL TRIAL: NCT00801034
Title: The Effects of Potassium on Physiological Variables in the Kidney and Cardiovascular Variables in Healthy Persons in a Double-blinded, Randomised, Placebo-controlled, Cross-over Study
Brief Title: The Effects of Potassium on Physiological and Cardiovascular Variables in Healthy Persons
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, professor, chief physician, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MED.RES.HOS.2008.01.SKM
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2011-12

CONDITIONS: Hypertension
Keywords: hypertension; potassium; blood pressure
MeSH Terms: conditions — Hypertension | interventions — Calcium; Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Calcium tablets
  Interventions: Drug: Calcium
- 2 (Active Comparator): Potassium tablets
  Interventions: Drug: Potassium

INTERVENTIONS:
Drug: Calcium — tablets, 1 tablet 2 times per day in 28 days
  Arms: 1
Drug: Potassium — Tablets, 5 tablets 2 times per day for 28 days
  Arms: 2

SUMMARY:
In humans living of fruit and vegetables, hypertension is rarely seen. We wish to study if the development of hypertension has a connection to our intake of potassium. We know that fruit and vegetables contain a lot of potassium and we will simulate this intake by giving healthy subjects potassium as tablets.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age 18-40 years old
* BMI 18, 5-30
* non-smoker

Exclusion Criteria:

* daily use of medicine
* alcohol or drugs
* desire to become pregnant
* not using safe anti-contraceptive
* abnormal results in the initial testing

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Effect on blood pressure | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of medical research, Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Matthesen SK, Larsen T, Vase H, Lauridsen TG, Pedersen EB. Effect of potassium supplementation on renal tubular function, ambulatory blood pressure and pulse wave velocity in healthy humans. Scand J Clin Lab Invest. 2012 Feb;72(1):78-86. doi: 10.3109/00365513.2011.635216. Epub 2011 Dec 12. PMID 22149452